CLINICAL TRIAL: NCT05329376
Title: Interactive Virtual Assistance for Self-Care Management and Mental Health Promotion in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidade Católica do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20220311
Record Dates: First submitted 2022-03-14; First posted 2022-04-15 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus, Type 2; Depression, Anxiety; Mental Health Disorder; Old Age; Debility
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Depression; Anxiety Disorders; Mental Disorders; Frailty

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): 12 weeks of daily interactions with Smart Speaker EchoDot 3rd Gen (Amazon Echo®).
  Interventions: Device: Smart Speaker Echo Dot
- Group B (Other): 12 weeks of maintenance of usual care.
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: Smart Speaker Echo Dot — Participants will receive the Smart Speaker EchoDot 3rd Gen (Amazon Echo®) device (i.e., Alexa) for home use, installed during a home visit following the study enrollment. In addition to the usual functionality of the system, the device will be programmed using a standard model developed by the research team, applied to each patient. The proposed model involves automatic interactions between the device and the patient, comprising:
  1. Medication reminders
  2. Glucose test reminders:
  3. Educational health tips
  4. Weekly educational podcasts
  5. Good morning and good night routine
  Arms: Group A
Other: Usual Care — Participants will maintain usual care during the study period and will receive a booklet with general advice following enrollment
  Arms: Group B

SUMMARY:
BACKGROUD: Health technology is an important tool in the aging process, which may improve the health condition and self-esteem of the elderly, in addition to offering new opportunities and challenges. In this scenario, the use of virtual interaction systems emerge as promising alternatives for the old adults, which often deals with the lack of social interaction, cognitive decline and decline in functional capacity, making the control of chronic diseases, such as diabetes, a challenge.

OBJECTIVES: This project aims to evaluate the effectiveness of using an interactive virtual assistance system in mental health parameters, glycemic profile and diabetes selfcare behavior in elderly people with diabetes.

METHODS: A randomized clinical trial is proposed, for an intervention that includes 3 months of use of the Smart Speaker Echo Dot system, programmed to provide reminders, stimulate treatment records and maintain healthy habits. Outcomes assessed will include parameters of mental health and diabetes control.

ELIGIBILITY:
Inclusion:

* Being 65 years of age or older;
* Having a diagnosis of type 2 diabetes;
* Residing in Porto Alegre or metropolitan region;
* Presenting availability of Wi-Fi connection at home; and
* Presenting availability to participate in the proposed face-to-face evaluation and accept receiving one visit for installation of the device.

Exclusion:

* Having an interactive virtual home assistance device at the time of enrollment;
* Having cognitive impairments or severe hearing impairments that prevent adequate interaction with outcome assessors and the application of follow-up questionnaires; or
* Residing in regions of difficult access.

Recruitment:

Study subjects will be recruited through two different strategies:

* Screening of records of the outpatients clinics of Hospital São Lucas (HSL)
* Social media advertising, specially in Instagram®

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 112 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Screening for depression, anxiety and common mental health disorders in elderly | Change from baseline to 12 weeks
  For mental health screening, the Self Report Questionnaire (SRQ 20) will be used, translated into Portuguese and validated for the Brazilian population. It is a questionnaire with 20 questions specially developed for the screening of depression, anxiety em common mental health disorders in the elderly. Higher scores indicating more mental distress.

SECONDARY OUTCOMES:
Glycemic control: glycated hemoglobin (HbA1c) assessment | Change from baseline to 12 weeks
  To assess glycemic control, the dosage of glycated hemoglobin (HbA1c) will be performed by high performance liquid chromatography, a measure that estimates the average glycemic control of the three months before the exam.
Variation in systolic blood pressure | Change from baseline to 12 weeks
  Systolic blood pressure assessment (mmHg)
Variation in diastolic blood pressure | Change from baseline to 12 weeks
  Diastolic blood pressure assessment (mmHg)
Variation in total cholesterol | Change from baseline to 12 weeks
  Total cholesterol (mg/dL)
Adherence parameters and self-care in the treatment of diabetes | Change from baseline to 12 weeks
  To assess adherence and self-care related to diabetes, the Self-Care Inventory Revised (SCI-R) questionnaire will be used, a version translated into Portuguese and validated for the Brazilian population. It is a questionnaire with 11 questions and answer options based on the 5-point Likert scale and which reflects the follow-up of treatment recommendations and lifestyle habits related to diabetes care in the2 months prior to the application. Higher scores reflect greater adherence and self-care.
Evaluation of quality of life | Change from baseline to 12 weeks
  Quality of Life will be assessed at baseline and after 12 weeks using the Short Form Health Survey (SF-36) questionnaire.
Perception of stress: | Change from baseline to 12 weeks
  Quality of Life will be assessed at baseline and after 12 weeks using the Perceived Stress Scale (PSS) questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Pontifícia Universidade Católica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Matzenbacher LS, da Costa FL, de Barros LGB, Gheno V, Maia IS, Blank LM, Brum MAB, Fontoura LF, Viola TW, Schwanke CHA, Gadonski G, Alessi J, Telo GH. Interactive Virtual Assistant for Health Promotion Among Older Adults With Type 2 Diabetes: The IVAM-ED Randomized Clinical Trial. JAMA Netw Open. 2026 Jan 2;9(1):e2553508. doi: 10.1001/jamanetworkopen.2025.53508. PMID 41575748
- [Derived] da Costa FL, Matzenbacher LS, Gheno V, Brum MAB, de Barros LGB, Maia IS, Blank LM, Fontoura LF, Alessi J, Telo GH. Interactive virtual assistance for mental health promotion and self-care management in elderly with type 2 diabetes (IVAM-ED): study protocol and statistical analysis plan for a randomized controlled trial. Trials. 2024 Mar 21;25(1):205. doi: 10.1186/s13063-024-08055-3. PMID 38515201